CLINICAL TRIAL: NCT06296121
Title: A Double-Blind, Randomized Clinical Study of the Efficacy and Safety of Monotherapy With BCD-264 and Darzalex® in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: A Study of the Efficacy and Safety of Monotherapy With BCD-264 and Darzalex in Subjects With Relapsed and Refractory Multiple Myeloma
Acronym: DARVIVA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-264-2
Record Dates: First submitted 2024-02-13; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-264 (Experimental): Blinded period: BCD-264 (daratumumab) will be administered intravenously once weekly for the first 8 weeks (Cycles 1 and 2), then once every two weeks for 16 weeks (Cycles 3, 4, 5 and 6). The total duration of the blinded treatment period is 6 cycles.
  Open-label period: starting from Day 1 of Cycle 7, the subjects will receive open-label BCD-264 once every 4 weeks
  Interventions: Drug: BCD-264
- Darzalex (Active Comparator): Blinded period: Darzalex (daratumumab) will be administered intravenously once weekly for the first 8 weeks (Cycles 1 and 2), then once every two weeks for 16 weeks (Cycles 3, 4, 5 and 6). The total duration of the blinded treatment period is 6 cycles.
  Open-label period: starting from Day 1 of Cycle 7, the subjects will receive open-label BCD-264 once every 4 weeks
  Interventions: Drug: Darzalex

INTERVENTIONS:
Drug: BCD-264 — IV, 16 mg/kg
  Other Names: daratumumab
  Arms: BCD-264
Drug: Darzalex — IV, 16 mg/kg
  Other Names: daratumumab
  Arms: Darzalex

SUMMARY:
The aim of this study is to confirm the comparability of the efficacy and safety profiles of BCD-264 and Darzalex as monotherapy for relapsed and refractory multiple myeloma in subjects previously treated with proteasome inhibitors and immunomodulatory drugs, and who had disease progression on prior therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Age ≥ 18 years at the time of signing of the informed consent form.
3. Documented diagnosis of multiple myeloma according to IMWG criteria
4. Measurable disease at screening:

   1. M-protein in serum ≥ 1.0 g/dL (10 g/L) or in 24-hour urine ≥ 200 mg; or
   2. light chain myeloma: serum "involved" FLC level ≥ 10 mg/dL (100 mg/L) and abnormal κ/λ FLC ratio .
5. At least a partial response according to IMWG criteria to at least 1 prior line of therapy.
6. Subjects with relapsed and refractory multiple myeloma who previously received therapy with proteasome inhibitors and immunomodulatory drugs, and who had disease progression on prior therapy
7. ECOG score 0-2.
8. Not pregnant and willing to use contraception.
9. Consent to bone marrow biopsy in the study.

Exclusion Criteria:

1. Prior treatment with daratumumab or other anti-CD38 therapy.
2. Prior treatment for multiple myeloma within 2 weeks or 5 half-lives before the date of randomization, except for a short course of glucocorticoids
3. Autologous hematopoietic stem cell transplantation within 12 weeks prior to the date of randomization.
4. Allogeneic hematopoietic stem cell transplantation, regardless of timing.
5. Scheduled hematopoietic stem cell transplantation prior to progressive disease during this study.
6. Plasma cell leukemia, POEMS syndrome or amyloidosis.
7. Waldenstrom macroglobulinemia or other concomitant diseases with hyperproduction of monoclonal IgM (M-protein) in the absence of clonal proliferation of plasma cells with lytic bone involvement.
8. A history of other malignancies within the last 5 years, with the exception of squamous cell and basal cell skin cancer, cervical, breast carcinoma in situ, or other non-invasive malignancies that, in the Investigator's opinion are considered to have been adequately treated and have a minimal risk of recurrence for 5 years.
9. Plasmapheresis within 28 days prior to randomization.
10. Clinical signs of meningeal involvement of multiple myeloma.
11. Pregnancy or breastfeeding, as well as planning pregnancy throughout the study and within 3 months after the last dose of daratumumab; for male subjects, planning to conceive a child throughout the study and within 3 months after the last dose of daratumumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall response rate according to IMWG (International Myeloma Working Group) criteria | up to 24 weeks

SECONDARY OUTCOMES:
Stringent complete response rate according to IMWG criteria | up to 3 years
Complete response (CR) rate according to IMWG criteria | up to 3 years
Very good partial response (VGPR) rate according to IMWG criteria | up to 3 years
Duration of response | up to 3 years
Progression-free survival | up to 3 years
Time to progression | up to 3 years
Time to response | up to 3 years
Overall survival | up to 3 years

OTHER OUTCOMES:
Incidence and characteristics of adverse events | up to 2 years
Proportion of subjects with BAbs/Nabs | up to 2 years
Time to BAb/NAb development | up to 2 years
AUC0-168 | up to Day 8 Cycle 1 (each cycle is 28 days)
AUC0-∞ | up to Day 15 Cycle 6 (each cycle is 28 days)
AUC0-336, ss | from Day 1 to Day 15 Cycle 6 (each cycle is 28 days)
Cmax | up to Day 15 Cycle 6 (each cycle is 28 days)
Cmax, ss | up to Day 15 Cycle 6 (each cycle is 28 days)
Tmax | up to Day 15 Cycle 6 (each cycle is 28 days)
T1/2 | up to Day 15 Cycle 6 (each cycle is 28 days)
Vd | up to Day 15 Cycle 6 (each cycle is 28 days)
Ctrough, ss | up to Day 15 Cycle 6 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (14):
- Russia (14):
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - Kuzbass Regional Clinical Hospital named after S.V. Belyaev, Kemerovo
  - Regional Clinical Hospital, Krasnoyarsk
  - Moscow City Clinical Hospital 52, Moscow
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Almazov National Medical Research Centre, Saint Petersburg
  - N.N. Petrov National Medicine Research Center of oncology, Saint Petersburg
  - Russian Research Institute of Hematology and Transfusiology of the Federal Medical and Biological Agency, Saint Petersburg
  - St Petersburg State I.P. Pavlov Medical University, Saint Petersburg
  - State budgetary healthcare institution Leningrad Regional Clinical Hospital, Saint Petersburg
  - Samara State Medical University, Samara
  - Oncological dispensary No. 2 of the Ministry of Health of the Krasnodar Territory, Sochi
  - Bashkir State Medical University, Ufa
  - Sverdlovsk Regional Clinical Hospital No. 1, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No